CLINICAL TRIAL: NCT06164964
Title: Study of Social Cognition Processes With Multimodal MRI on Healthy Adult Patients.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: SOCIOCOGN
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Social Cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: study of higher cognitive functions — General objective: increase knowledge about neural correlates:
  of the cognitive processing of stimuli of a social nature; of decision-making processes in the context of individual choice; of the influence of the social context on individual decision-making processes.

SUMMARY:
The study of higher cognitive functions (learning, memory, language, reasoning, decision making) in humans constitutes an interdisciplinary field, which combines neurobiological and neurological, neuropsychological, as well as linguistic and artificial intelligence skills. Historically, the study of patients with cerebrovascular lesions or brain pathologies associated with primary and/or cognitive deficits has produced fundamental knowledge in this area. The development of modern non-invasive investigation techniques of the human brain - such as Structural Magnetic Resonance Imaging (MRI), Diffusion Tensor Imaging, Functional Magnetic Resonance Imaging (fMRI), Positron emission (PET), the study of event-related electrophysiological potentials (ERP) or magneto-encephalography (MEG) - has made it possible to carry out similar studies on healthy subjects, as well as the in-vivo analysis of adaptive and plastic mechanisms of the human brain. Recently, the interest of cognitive neuroscience - this is the name taken by this vast interdisciplinary sector which aims to understand the neural mechanisms underlying human cognitive processes - has been oriented towards the study of decision making in social contexts. Knowledge of the mechanisms underlying these processes is fundamental for the most complete description of the biological bases of human behavior and above all for the optimal development of treatments for brain pathologies, whether surgical, pharmacological or rehabilitation in general.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years old; Monolingual native speakers of Italian; Absence of neurological or psychiatric pathologies that could interfere with carrying out the exam.

Exclusion Criteria:

* Clinical and/or anamnestic evidence of significant neuropsychiatric or systemic pathologies; Previous head trauma with loss of consciousness

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Behavioral study with neuro-anatomical functional correlates consisting of cognitive activation experiments during functional magnetic resonance imaging, with observation of images of a social nature and decision making in an individual or social context.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-04-22 (Actual); Primary Completion 2010-10-28 (Actual); Study Completion 2010-10-28 (Actual)

PRIMARY OUTCOMES:
behavioral study with neuroanatomical functional correlates consisting of cognitive activation experiments during functional magnetic resonance imaging | 1 year

IPD SHARING:
Plan to Share IPD: No